CLINICAL TRIAL: NCT05967039
Title: Evaluation of Lung Function, Lung Ultrasound and Functional Capacity in Long-COVID Patients Who Underwent Physical Therapy
Brief Title: Assessment of Functional Capacity in Long-COVID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Other Study IDs: 30135320.0.0000.5259
Record Dates: First submitted 2023-07-03; First posted 2023-08-01 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Post-COVID-19 Syndrome; Long COVID
Keywords: Functional capacity;; Six-minute walk test;; Spirometry;; Oscillometry;; Lung Ultrasound;; Ventilometry;
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: This is a control group of individuals who were diagnosed with post-COVID-19 syndrome but did not underwent Physiotherapy.
  Interventions: Other: Physiotherapy
- Intervention: This is an intervention group of individuals who were diagnosed with post-COVID-19 syndrome and underwent Physiotherapy
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Physiotherapy in respiratory rehabilitation

SUMMARY:
A paucity of prognostic studies in patients with post-COVID-19 syndrome (long-COVID) shows the need to identify the main effects on functional capacity in the short and medium term. In this regard, the evaluation of lung function, lung structure and functional capacity in long-COVID patients is essential to estimate the impact of the disease. This retrospective observational study aims to compare functional capacity, lung function, and lung ultrasound findings in patients who underwent physical therapy to those who did not.

DETAILED DESCRIPTION:
Introduction: The pandemic caused by the Severe acute respiratory syndrome by coronavirus 2 (SARS-CoV-2) has been presented as a one of the greatest health challenges on a global scale at the beginning of this millennium. Many patients need physical therapy in their recovery process. A paucity of prognostic studies in patients with long-COVID shows the need to identify the main repercussions on functional capacity in the short and medium term. In this regard, the evaluation of lung function, lung structure and functional capacity in long-COVID patients is essential to estimate the impact of the disease.

Objective: The present study aims to compare functional capacity, lung function, and lung ultrasound findings between patients diagnosed with long-COVID who underwent physical therapy to those who did not.

Methods: This is a retrospective observational study with quantitative data analysis. The study will be carried out at the Pulmonary Function Laboratory of the Policlínica Universitária Piquet Carneiro, from the State University of Rio de Janeiro. First, a clinical evaluation will be performed. In the survey, it will be asked whether the patient had undergone physical therapy treatment, so they can be allocated in the control or intervention group. After that, they will answer to the Post-COVID-19 Functional Status Scale (PCFS), a tool to measure functional status over time after COVID-19. Then, patients will have their lung function evaluated through spirometry and impulse oscillometry (IOS). In addition, lung ultrasound (LUS) images will be analyzed. And their functional capacity will be assessed using the six-minute walk test (6MWT) coupled to pulmonary ventilation measurement using Spiropalm® (Spiropalm 6MWT, Cosmed, Rome, Italy).

It is expected that understanding the consequences of long-COVID on pulmonary ventilation can help to design therapeutic strategies in rehabilitation services.

ELIGIBILITY:
Inclusion Criteria:

Individuals with an established diagnosis of COVID-19 (RT-PCR) who required hospitalization or not, regardless of whether or not they were treated in the ICU.

Exclusion Criteria:

Patients unable to perform the tests. Patients with musculoskeletal disorders not associated with COVID-19. Patients with lung, heart or cerebrovascular diseases not associated with COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with long-COVID-19 syndrome
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test coupled into the measurement of pulmonary ventilation | October 2023
  The individuals will undergo the six-minute walk test coupled to the measurement of ventilation using equipment using a face mask with monitoring of ventilatory variables and vital signs on a 30-meter track where the purpose is to assess the functional capacity

SECONDARY OUTCOMES:
Impulse oscillometry | October 2023
  The IOS will be performed using an impulse oscillometer (Quark i2m, Cosmed, Rome Italy). During the IOS assessment, participants will be guided to stay seated, keeping the head in a neutral position, with manual support on the cheeks and with the nostrils occluded by a clip and then they will breathe usually for 40 seconds (ALBUQUERQUE et al., 2015). The values of acceptable minimum coherence will be ≥0.9 Hz. The following resistive and reactive parameters were evaluated: Rsr at 4 Hz (R4), 6 Hz (R6), 10 Hz (R10) and 20 Hz (R20); average resistance between 4-20 Hz (Rm); heterogeneity of resistance between R4 and R20 (R4-R20); resonant frequency (Fres); and area under reactance curve (AX). The values of R4, R6, R10 and R20 will be considered 34 abnormal when ≥150% of predicted (OOSTVEEN et al., 2013). A change in Fres and AX will be considered when >12 Hz and >3.60 cm H2O/L/s, respectively (BERGER et al., 2013).
Spirometry | October 2023
  It is a procedure that allows the diagnosis of ventilatory disorders and is capable of measuring the patient's pulmonary function - evaluating the volume and velocity of the air blown. It is done with the aid of a device, the spirometer. The patient breathes into this device and internal sensors measure the amount of air and air movement in the lungs.
Lung ultrasound | October 2023
  Participants will perform the LUS on Aplio XG equipment Aplio XG (Toshiba Medical Systems, Tokyo, Japan) coupled to a linear transducer 7.5-10 megahertz (MHz) multi-frequency transducer or a 3.5-5 MHz convex transducer in B. All USP evaluations will be performed by the authors who, although not whether they are radiologists, they are all employees of Policlínica Piquet Carneiro and have at least least 9 years of USP experience at the participant screening site. All USP assessments will be performed by 2 examiners and, when disagreement between them will be resolved through collective discussion. With participants in a seated position, the capture of USP signals will be done in 6 areas of each hemithorax as follows (SOUMMER et al., 2012): two anterior, two side and two back. In the evaluation of the pathological signs of USP, the investigators will search for B lines >2, coalescing B lines, and subpleural consolidations (MAFORT et al., 2021).
Functional Status scale PCFS | October 2023
  The Post-COVID-19 Functional Status scale: a tool to measure functional status over time after COVID-19, being a self-administered questionnaire for the patient who will be informed: how much are you currently affected in your daily life by COVID 19? The patient will indicate in a classification from 0 to 4 their degree of functional status

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Agnaldo José Lopes, Rio de Janeiro
  - Centro Universitario Augusto Motta, Rio de Janeiro

REFERENCES:
- [Background] Ahmad FB, Cisewski JA, Minino A, Anderson RN. Provisional Mortality Data - United States, 2020. MMWR Morb Mortal Wkly Rep. 2021 Apr 9;70(14):519-522. doi: 10.15585/mmwr.mm7014e1. PMID 33830988
- [Background] Al-Ani F, Chehade S, Lazo-Langner A. Thrombosis risk associated with COVID-19 infection. A scoping review. Thromb Res. 2020 Aug;192:152-160. doi: 10.1016/j.thromres.2020.05.039. Epub 2020 May 27. PMID 32485418
- [Background] Albuquerque CG, Andrade FM, Rocha MA, Oliveira AF, Ladosky W, Victor EG, Rizzo JA. Determining respiratory system resistance and reactance by impulse oscillometry in obese individuals. J Bras Pneumol. 2015 Sep-Oct;41(5):422-6. doi: 10.1590/S1806-37132015000004517. PMID 26578133
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Andersen KG, Rambaut A, Lipkin WI, Holmes EC, Garry RF. The proximal origin of SARS-CoV-2. Nat Med. 2020 Apr;26(4):450-452. doi: 10.1038/s41591-020-0820-9. No abstract available. PMID 32284615
- [Background] Bahl P, Doolan C, de Silva C, Chughtai AA, Bourouiba L, MacIntyre CR. Airborne or Droplet Precautions for Health Workers Treating Coronavirus Disease 2019? J Infect Dis. 2022 May 4;225(9):1561-1568. doi: 10.1093/infdis/jiaa189. PMID 32301491
- [Background] Bansal M. Cardiovascular disease and COVID-19. Diabetes Metab Syndr. 2020 May-Jun;14(3):247-250. doi: 10.1016/j.dsx.2020.03.013. Epub 2020 Mar 25. PMID 32247212
- [Background] Barker-Davies RM, O'Sullivan O, Senaratne KPP, Baker P, Cranley M, Dharm-Datta S, Ellis H, Goodall D, Gough M, Lewis S, Norman J, Papadopoulou T, Roscoe D, Sherwood D, Turner P, Walker T, Mistlin A, Phillip R, Nicol AM, Bennett AN, Bahadur S. The Stanford Hall consensus statement for post-COVID-19 rehabilitation. Br J Sports Med. 2020 Aug;54(16):949-959. doi: 10.1136/bjsports-2020-102596. Epub 2020 May 31. PMID 32475821
- [Background] Beraldo GL, Fonseca EKUN, Yokoo P, Matos MJR, Rosa MEE, Silva MMA, Chate RC, Shoji H, Ishikawa WY. Novel coronavirus pneumonia and acute pulmonary thromboembolism: casualty or causality? Einstein (Sao Paulo). 2020 Jun 3;18:eAI5750. doi: 10.31744/einstein_journal/2020AI5750. eCollection 2020. No abstract available. PMID 32520072
- [Background] Berger KI, Reibman J, Oppenheimer BW, Vlahos I, Harrison D, Goldring RM. Lessons from the World Trade Center disaster: airway disease presenting as restrictive dysfunction. Chest. 2013 Jul;144(1):249-257. doi: 10.1378/chest.12-1411. PMID 23392588
- [Background] Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID 32227758
- [Background] Biryukov J, Boydston JA, Dunning RA, Yeager JJ, Wood S, Ferris A, Miller D, Weaver W, Zeitouni NE, Freeburger D, Dabisch P, Wahl V, Hevey MC, Altamura LA. SARS-CoV-2 is rapidly inactivated at high temperature. Environ Chem Lett. 2021;19(2):1773-1777. doi: 10.1007/s10311-021-01187-x. Epub 2021 Feb 3. PMID 33551702
- [Background] Buonsenso D, Sali M, Pata D, De Rose C, Sanguinetti M, Valentini P, Delogu G. Children and COVID-19: Microbiological and immunological insights. Pediatr Pulmonol. 2020 Oct;55(10):2547-2555. doi: 10.1002/ppul.24978. Epub 2020 Jul 30. PMID 32710652
- [Background] Butzko RP, Sotolongo AM, Helmer DA, Klein-Adams JC, Osinubi OY, Berman AR, Ortiz-Pacheco R, Falvo MJ. Forced oscillation technique in veterans with preserved spirometry and chronic respiratory symptoms. Respir Physiol Neurobiol. 2019 Feb;260:8-16. doi: 10.1016/j.resp.2018.11.012. Epub 2018 Nov 30. PMID 30508589
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Chan JF, To KK, Tse H, Jin DY, Yuen KY. Interspecies transmission and emergence of novel viruses: lessons from bats and birds. Trends Microbiol. 2013 Oct;21(10):544-55. doi: 10.1016/j.tim.2013.05.005. Epub 2013 Jun 14. PMID 23770275
- [Background] Colavita F, Lapa D, Carletti F, Lalle E, Bordi L, Marsella P, Nicastri E, Bevilacqua N, Giancola ML, Corpolongo A, Ippolito G, Capobianchi MR, Castilletti C. SARS-CoV-2 Isolation From Ocular Secretions of a Patient With COVID-19 in Italy With Prolonged Viral RNA Detection. Ann Intern Med. 2020 Aug 4;173(3):242-243. doi: 10.7326/M20-1176. Epub 2020 Apr 17. No abstract available. PMID 32302380
- [Background] Costa IBSDS, Bittar CS, Rizk SI, Araujo Filho AE, Santos KAQ, Machado TIV, Andrade FTA, Gonzalez TB, Arevalo ANG, Almeida JP, Bacal F, Oliveira GMM, Lacerda MVG, Barberato SH, Chagas ACP, Rochitte CE, Ramires JAF, Kalil Filho R, Hajjar LA. The Heart and COVID-19: What Cardiologists Need to Know. Arq Bras Cardiol. 2020 May 11;114(5):805-816. doi: 10.36660/abc.20200279. English, Portuguese. PMID 32401847
- [Background] Demeco A, Marotta N, Barletta M, Pino I, Marinaro C, Petraroli A, Moggio L, Ammendolia A. Rehabilitation of patients post-COVID-19 infection: a literature review. J Int Med Res. 2020 Aug;48(8):300060520948382. doi: 10.1177/0300060520948382. PMID 32840156
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Gonzalez J, Zuil M, Benitez ID, de Gonzalo-Calvo D, Aguilar M, Santisteve S, Vaca R, Minguez O, Seck F, Torres G, de Batlle J, Gomez S, Barril S, Moncusi-Moix A, Monge A, Gort-Paniello C, Ferrer R, Ceccato A, Fernandez L, Motos A, Riera J, Menendez R, Garcia-Gasulla D, Penuelas O, Labarca G, Caballero J, Barbera C, Torres A, Barbe F. One Year Overview and Follow-Up in a Post-COVID Consultation of Critically Ill Patients. Front Med (Lausanne). 2022 Jul 14;9:897990. doi: 10.3389/fmed.2022.897990. eCollection 2022. PMID 35911414
- [Background] Pitta F, Troosters T, Spruit MA, Probst VS, Decramer M, Gosselink R. Characteristics of physical activities in daily life in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 May 1;171(9):972-7. doi: 10.1164/rccm.200407-855OC. Epub 2005 Jan 21. PMID 15665324
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Guler MA, Guler K, Guneser Gulec M, Ozdoglar E. Working From Home During a Pandemic: Investigation of the Impact of COVID-19 on Employee Health and Productivity. J Occup Environ Med. 2021 Sep 1;63(9):731-741. doi: 10.1097/JOM.0000000000002277. PMID 34091577
- [Background] Hui DS, Wong KT, Ko FW, Tam LS, Chan DP, Woo J, Sung JJ. The 1-year impact of severe acute respiratory syndrome on pulmonary function, exercise capacity, and quality of life in a cohort of survivors. Chest. 2005 Oct;128(4):2247-61. doi: 10.1378/chest.128.4.2247. PMID 16236881
- [Background] Hussain A, Baleanu D, Adeel M. Existence of solution and stability for the fractional order novel coronavirus (nCoV-2019) model. Adv Differ Equ. 2020;2020(1):384. doi: 10.1186/s13662-020-02845-0. Epub 2020 Jul 25. PMID 32834817
- [Background] Ianniello S, Di Giacomo V, Sessa B, Miele V. First-line sonographic diagnosis of pneumothorax in major trauma: accuracy of e-FAST and comparison with multidetector computed tomography. Radiol Med. 2014 Sep;119(9):674-80. doi: 10.1007/s11547-014-0384-1. Epub 2014 Jan 28. PMID 24469989
- [Background] van Kampen JJA, van de Vijver DAMC, Fraaij PLA, Haagmans BL, Lamers MM, Okba N, van den Akker JPC, Endeman H, Gommers DAMPJ, Cornelissen JJ, Hoek RAS, van der Eerden MM, Hesselink DA, Metselaar HJ, Verbon A, de Steenwinkel JEM, Aron GI, van Gorp ECM, van Boheemen S, Voermans JC, Boucher CAB, Molenkamp R, Koopmans MPG, Geurtsvankessel C, van der Eijk AA. Duration and key determinants of infectious virus shedding in hospitalized patients with coronavirus disease-2019 (COVID-19). Nat Commun. 2021 Jan 11;12(1):267. doi: 10.1038/s41467-020-20568-4. PMID 33431879
- [Background] Kang N, Shin SH, Gu S, Kang D, Cho J, Jeong HJ, Suh GY, Lee H, Park HY. The impact of low forced vital capacity on behavior restrictions in a population with airflow obstruction. J Thorac Dis. 2019 Apr;11(4):1316-1324. doi: 10.21037/jtd.2019.03.77. PMID 31179073
- [Background] Kanne JP, Little BP, Chung JH, Elicker BM, Ketai LH. Essentials for Radiologists on COVID-19: An Update-Radiology Scientific Expert Panel. Radiology. 2020 Aug;296(2):E113-E114. doi: 10.1148/radiol.2020200527. Epub 2020 Feb 27. No abstract available. PMID 32105562
- [Background] Lopes AJ, de Menezes SL, Dias CM, de Oliveira JF, Mainenti MR, Guimaraes FS. Comparison between cardiopulmonary exercise testing parameters and computed tomography findings in patients with thoracic sarcoidosis. Lung. 2011 Oct;189(5):425-31. doi: 10.1007/s00408-011-9316-1. Epub 2011 Aug 20. PMID 21858420
- [Background] Lopes AJ, Mafort TT, da Cal MS, Monnerat LB, Litrento PF, Ramos I, de Oliveira RFJ, da Costa CH, Rufino R. Impulse Oscillometry Findings and Their Associations With Lung Ultrasound Signs in COVID-19 Survivors. Respir Care. 2021 Nov;66(11):1691-1698. doi: 10.4187/respcare.09193. Epub 2021 Sep 7. PMID 34493607
- [Background] Lutchmansingh DD, Knauert MP, Antin-Ozerkis DE, Chupp G, Cohn L, Dela Cruz CS, Ferrante LE, Herzog EL, Koff J, Rochester CL, Ryu C, Singh I, Tickoo M, Winks V, Gulati M, Possick JD. A Clinic Blueprint for Post-Coronavirus Disease 2019 RECOVERY: Learning From the Past, Looking to the Future. Chest. 2021 Mar;159(3):949-958. doi: 10.1016/j.chest.2020.10.067. Epub 2020 Nov 4. PMID 33159907
- [Background] Mafort TT, Rufino R, da Costa CH, da Cal MS, Monnerat LB, Litrento PF, Parra LLZ, Marinho ASES, Lopes AJ. One-month outcomes of patients with SARS-CoV-2 infection and their relationships with lung ultrasound signs. Ultrasound J. 2021 Apr 9;13(1):19. doi: 10.1186/s13089-021-00223-9. PMID 33835273
- [Background] Mitchell JH, Levine BD, McGuire DK. The Dallas Bed Rest and Training Study: Revisited After 50 Years. Circulation. 2019 Oct 15;140(16):1293-1295. doi: 10.1161/CIRCULATIONAHA.119.041046. Epub 2019 Oct 14. No abstract available. PMID 31609661
- [Background] NEWS MEDICAL. Spiropalm Handheld Spirometer from COSMED. Medical Devices, Spirometers, 2022. Disponível em: <https://www.news- medical.net/Spiropalm-Handheld-Spirometer-from-COSMED>. Acesso em 10 de novembro de 2022
- [Background] Ngai JC, Ko FW, Ng SS, To KW, Tong M, Hui DS. The long-term impact of severe acute respiratory syndrome on pulmonary function, exercise capacity and health status. Respirology. 2010 Apr;15(3):543-50. doi: 10.1111/j.1440-1843.2010.01720.x. Epub 2010 Mar 19. PMID 20337995
- [Background] Onder G, Rezza G, Brusaferro S. Case-Fatality Rate and Characteristics of Patients Dying in Relation to COVID-19 in Italy. JAMA. 2020 May 12;323(18):1775-1776. doi: 10.1001/jama.2020.4683. No abstract available. PMID 32203977
- [Background] Oostveen E, Boda K, van der Grinten CP, James AL, Young S, Nieland H, Hantos Z. Respiratory impedance in healthy subjects: baseline values and bronchodilator response. Eur Respir J. 2013 Dec;42(6):1513-23. doi: 10.1183/09031936.00126212. Epub 2013 Apr 18. PMID 23598954
- [Background] Oreshkova N, Molenaar RJ, Vreman S, Harders F, Oude Munnink BB, Hakze-van der Honing RW, Gerhards N, Tolsma P, Bouwstra R, Sikkema RS, Tacken MG, de Rooij MM, Weesendorp E, Engelsma MY, Bruschke CJ, Smit LA, Koopmans M, van der Poel WH, Stegeman A. SARS-CoV-2 infection in farmed minks, the Netherlands, April and May 2020. Euro Surveill. 2020 Jun;25(23):2001005. doi: 10.2807/1560-7917.ES.2020.25.23.2001005. PMID 32553059
- [Background] Pasnick S, Carlos WG, Dela Cruz CS, Gross JE, Garrison G, Jamil S. SARS-CoV-2 Transmission and the Risk of Aerosol Generating Procedures. Am J Respir Crit Care Med. 2020 Jun 30. doi: 10.1164/rccm.2020C11. Online ahead of print. No abstract available. PMID 32603230
- [Background] Peng X, Xu X, Li Y, Cheng L, Zhou X, Ren B. Transmission routes of 2019-nCoV and controls in dental practice. Int J Oral Sci. 2020 Mar 3;12(1):9. doi: 10.1038/s41368-020-0075-9. PMID 32127517
- [Background] Sant'Anna M Jr, Carvalhal RF, Oliveira FDFB, Zin WA, Lopes AJ, Lugon JR, Guimaraes FS. Respiratory mechanics of patients with morbid obesity. J Bras Pneumol. 2019 Oct 17;45(5):e20180311. doi: 10.1590/1806-3713/e20180311. eCollection 2019. PMID 31644708
- [Background] Savioli F, Rocha LL. Coagulation profile in severe COVID-19 patients: what do we know so far? Rev Bras Ter Intensiva. 2020 Jun;32(2):197-199. doi: 10.5935/0103-507x.20200031. Epub 2020 Jun 24. No abstract available. PMID 32667446
- [Background] Sibila M, Guevara G, Cuadrado R, Pleguezuelos P, Perez D, Perez de Rozas A, Huerta E, Llorens A, Valero O, Perez M, Lopez C, Krejci R, Segales J. Comparison of Mycoplasma hyopneumoniae and porcine circovirus 2 commercial vaccines efficacy when applied separate or combined under experimental conditions. Porcine Health Manag. 2020 May 4;6:11. doi: 10.1186/s40813-020-00148-0. eCollection 2020. PMID 32391165
- [Background] Soldati G, Smargiassi A, Inchingolo R, Buonsenso D, Perrone T, Briganti DF, Perlini S, Torri E, Mariani A, Mossolani EE, Tursi F, Mento F, Demi L. Proposal for International Standardization of the Use of Lung Ultrasound for Patients With COVID-19: A Simple, Quantitative, Reproducible Method. J Ultrasound Med. 2020 Jul;39(7):1413-1419. doi: 10.1002/jum.15285. Epub 2020 Apr 13. PMID 32227492
- [Background] Sutton D, Fuchs K, D'Alton M, Goffman D. Universal Screening for SARS-CoV-2 in Women Admitted for Delivery. N Engl J Med. 2020 May 28;382(22):2163-2164. doi: 10.1056/NEJMc2009316. Epub 2020 Apr 13. No abstract available. PMID 32283004
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Thachil J, Tang N, Gando S, Falanga A, Cattaneo M, Levi M, Clark C, Iba T. ISTH interim guidance on recognition and management of coagulopathy in COVID-19. J Thromb Haemost. 2020 May;18(5):1023-1026. doi: 10.1111/jth.14810. Epub 2020 Apr 27. No abstract available. PMID 32338827
- [Background] Torres-Castro R, Vasconcello-Castillo L, Alsina-Restoy X, Solis-Navarro L, Burgos F, Puppo H, Vilaro J. Respiratory function in patients post-infection by COVID-19: a systematic review and meta-analysis. Pulmonology. 2021 Jul-Aug;27(4):328-337. doi: 10.1016/j.pulmoe.2020.10.013. Epub 2020 Nov 25. PMID 33262076
- [Background] Caglar Tosun BN, Zeren M, Barlik M, Demir E, Gulen F. Investigation of dynamic hyperinflation and its relationship with exercise capacity in children with bronchiectasis. Pediatr Pulmonol. 2022 Sep;57(9):2218-2226. doi: 10.1002/ppul.26028. Epub 2022 Jun 14. PMID 35666051
- [Background] Williams FMK, Muirhead N, Pariante C. Covid-19 and chronic fatigue. BMJ. 2020 Jul 30;370:m2922. doi: 10.1136/bmj.m2922. No abstract available. PMID 32732337
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Ye Z, Wang Y, Colunga-Lozano LE, Prasad M, Tangamornsuksan W, Rochwerg B, Yao L, Motaghi S, Couban RJ, Ghadimi M, Bala MM, Gomaa H, Fang F, Xiao Y, Guyatt GH. Efficacy and safety of corticosteroids in COVID-19 based on evidence for COVID-19, other coronavirus infections, influenza, community-acquired pneumonia and acute respiratory distress syndrome: a systematic review and meta-analysis. CMAJ. 2020 Jul 6;192(27):E756-E767. doi: 10.1503/cmaj.200645. Epub 2020 May 14. PMID 32409522
- [Background] Zhang T, Wu Q, Zhang Z. Probable Pangolin Origin of SARS-CoV-2 Associated with the COVID-19 Outbreak. Curr Biol. 2020 Apr 6;30(7):1346-1351.e2. doi: 10.1016/j.cub.2020.03.022. Epub 2020 Mar 19. PMID 32197085
- [Background] Du Z, Xu X, Wu Y, Wang L, Cowling BJ, Meyers LA. Serial Interval of COVID-19 among Publicly Reported Confirmed Cases. Emerg Infect Dis. 2020 Jun;26(6):1341-1343. doi: 10.3201/eid2606.200357. Epub 2020 Jun 17. PMID 32191173